CLINICAL TRIAL: NCT03623152
Title: Colorectal Neoplasia and Microbiota: Does Left Equal Right?
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Joseph JY SUNG, Professor, Chinese University of Hong Kong
Other Study IDs: CRC MIC L&R
Record Dates: First submitted 2018-08-07; First posted 2018-08-09 (Actual); Last update posted 2019-07-24 (Actual); Status verified 2019-07

CONDITIONS: Colo-rectal Cancer
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Colonic biopsies from each site, stool and blood will be collected
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Many studies, including our own, have shown that colorectal cancer (CRC) is related to changes in the microbiome of the colon. However, there are limitations in most studies and questions remained unanswered. Some early data showing that the microbiome in the left vs right colon are different.

The aim of this study is to investigate the microbiome (including bacteriome, virome, and fungome) of adenoma/CRC comparing the left (distal to splenic flexure) vs right side (proximal to splenic flexure) of the colon.

DETAILED DESCRIPTION:
1. Many studies, including our own, have shown that colorectal cancer (CRC) is related to changes in the microbiome of the colon

   1. Certain bacterial phyla are more frequently presented in CRC
   2. Bacterial diversity is reduced in CRC
   3. Co-occurrence of bacterial phyla and exclusion are identified in CRC
   4. Besides bacteriome, viromes have been found associated with CRC
   5. These changes in the pattern may actually be used for diagnosis and prognosticate purposes.
2. However, there are limitations in most studies and questions remained unanswered

   1. Most studies used stool sample and data of tissue (tumor and adjacent normal tissues) may not be available
   2. Most studies take adenoma and CRC as one condition, without differentiating the findings according to tumor location
   3. Most studies have separate bacteria, virus and fungi. There is a lack of data on their interaction
   4. Most studies have identified either microbiome without correlating them with the genomic of the host
3. We know that not all CRC are the same. It has been known that rectal and colonic cancer are not the same. Furthermore, proximal (right) CRC and distal (left) CRC may not be the same.

   1. Studies have shown compare to L-CRC, patients with R-CRC are older, more female (Iaocopetta B et al. Int J Cancer 2002)
   2. Studies have also shown that the genomic make up of L-CRC and R-CRC are different. R-CRC are more likely to have family cancer syndrome (HNPCC), mostly diploid, less frequent to have loss heterozygosity, less TP53 mutations and more MSI and CIMP, and the gene expression are different (Glebov et al. Cancer Epi, Biomarker and Prevention 2003)
   3. The response to therapy might also be different in the L-CRC compare to R-CRC
   4. Recent studies show that the clinico-pathological and molecular features of early-onset (<50 years) CRC varies according to tumor location. (Peres J et al. Am J Cancer Res 2015). In the R-CRC in this group, germline mutation is more common (MLH1, MSH2, MSH6, PMS2 and EPCAM). Adenomas tend to be larger, flatter and more likely to have high-grade dysplasia and villous histology
   5. Recent studies have also shown that the clinic-pathological and molecular feature of in the late-onset CRC (70-80 years) varies with tumor location (Brandariz et al. Oncotarget 2018). There are more sporadic MSI, more BRAF mutation and the adenoma/CRC are likely to be mucinous.
4. Studies comparing the microbiome of L-CRC vs R-CRC has not been many. There is some early data showing that the microbiome in the left vs right colon are different.

The aim of this study is to investigate the microbiome (including bacteriome, virome, and fungome) of adenoma/CRC comparing the left (distal to splenic flexure) vs right side (proximal to splenic flexure) of the colon.

ELIGIBILITY:
Inclusion Criteria:

1. >18 years of age, with the informed consent of the study-specific colonoscopy examination method and samples collection
2. have an indication for a scheduled colonoscopy, either as an investigation of colorectal symptom or as part of a CRC screening
3. for those who are known to have either adenoma or CRC, colonoscopy is arranged for endoscopic submucosal dissection (ESD) or endoscopic mucosectomy (EMR)

Exclusion Criteria:

a. known history of coagulopathy b. recently on antithrombotics or antiplatelets c. recently on antibiotics, prebiotics, probiotics and symbiotics d. anticipated prolonged standard colonoscopy procedure at endoscopist's discretion e. consent cannot be obtained

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients have scheduled colonoscopy
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2018-08-07 (Actual); Primary Completion 2019-09-06 (Estimated); Study Completion 2019-10-06 (Estimated)

PRIMARY OUTCOMES:
Descriptive statistics will be used for demographics data | All biological samples will be stored for a maximum of 10 years
  Since the sample size is small, non-parametric chi-square test or Mann-Whitney tests will be used for the comparison of the clinical data between the cases with adenoma or CRC on the right and left side colon.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph JY Sung, Principal Investigator — Chinese Univeristy of Hong Kong
Locations (1):
- Endoscopy Center, Prince of Wales Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided